CLINICAL TRIAL: NCT05406843
Title: Postoperative Cognitive Dysfunction in Participants Undergoing Open Heart Surgery
Brief Title: Postoperative Cognitive Dysfunction in Heart Surgery
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Huri Yeşildal, Assistant, Kocaeli University
Other Study IDs: Observational
Record Dates: First submitted 2021-02-18; First posted 2022-06-07 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: COGNITIVE DYSFUNCTİON; HEART SURGERY; POSTOPERATIVE DELIRIUM
MeSH Terms: conditions — Postoperative Cognitive Complications; Cognition Disorders; Emergence Delirium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preoperative cognitive status of participants undergoing open heart surgery: Detection of postoperative cognitive impairment is difficult and it starts with testing in the preoperative period.
  In this study, it was aimed to determine postoperative cognitive impairment by comparing cognitive functions by using Minimental status test in the preoperative period in participants scheduled for open heart surgery for one year. It was planned to compare the obtained data in terms of participants undergoing valve and coronary bypass surgery, age, gender, diabetes, kidney disease, chronic obstructive pulmonary disease (COPD), surgical characteristics, bypass time, and crossclamping time.
  Interventions: Other: Preoperative cognitive functions of participants undergoing open heart surgery
- Postoperative cognitive status of participants undergoing open heart surgery: Detection of postoperative cognitive impairment is difficult and it starts with testing in the preoperative period. In this study, it was aimed to determine the postoperative cognitive impairment by comparing it with the cognitive functions in the preoperative period using the Minimental status test in the postoperative period in participants scheduled for open heart surgery for a year. It was planned to compare the obtained data in terms of participants undergoing valve and coronary bypass surgery, age, gender, diabetes, kidney disease, chronic obstructive pulmonary disease (COPD), surgical characteristics, bypass time, and crossclamping time.
  Interventions: Other: Postoperative cognitive functions of particiants undergoing open heart surgery

INTERVENTIONS:
Other: Preoperative cognitive functions of participants undergoing open heart surgery — Surgery times and cross-clamping times of the participants who will undergo open heart surgery were recorded.
  Groups: Preoperative cognitive status of participants undergoing open heart surgery
Other: Postoperative cognitive functions of particiants undergoing open heart surgery — Changes in mini mental test scores were recorded in the postoperative period.
  Groups: Postoperative cognitive status of participants undergoing open heart surgery

SUMMARY:
To determine the rate of Postoperative Cognitive Dysfunction (POCD) in the early and late postoperative periods by comparing the preop and postop period mini mental status tests in participants undergoing open heart surgery, and to compare the results of the investgators clinic with the world literature.

DETAILED DESCRIPTION:
Postoperative delirium (POD) and Cognitive Dysfunction (POCD) are changes in mental status, especially in the geriatric surgery population.Unlike other forms of delirium, POD results in early full recovery.Postoperative Cognitive Dysfunction (POCD) is more difficult to define and implies temporal consciousness impairment associated with surgery.

While the diagnosis of delirium requires the detection of symptoms, the diagnosis of POCD requires preoperative neuropsychological testing and determining how much reduction will mean cognitive dysfunction. Postoperative delirium management is complex and requires multiple strategies. Methods of treating and preventing POCD are still uncertain.It is known that POCD is most commonly seen in patients undergoing open heart surgery.In this study, the investigators aim is to evaluate whether there is any change in cognitive status in the postoperative period compared to the preoperative period of participants who will undergo open heart surgery due to valve pathology or coronary stenosis.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 age
* American Society of Anesthesiologists (ASA) II-III

Exclusion Criteria:

* >75 age
* <18 age
* Patients who died within 48 hours after the operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A study was planned on 140 patients undergoing open heart surgery.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of postoperative cognitive functions in participants undergoing open heart surgery. | 1 year
  The aim is to understand whether there is a loss of cognitive functions in the postoperative period, according to the preoperative periods, by testing the participants with open heart surgery on the 3rd day, 7th day, and 2nd month after the surgery.

SECONDARY OUTCOMES:
Comparison with the literature. | 1 year
  Comparison of the results in the investigators clinic with the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Tülay Çardaközü, Study Director — Kocaeli University
Locations (1):
- Kocaeli Üniversitesi Tıp Fakültesi Hastanesi, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected individual participant data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: The study results can be accessed by anyone who is a healthcare worker.